CLINICAL TRIAL: NCT03787576
Title: Relationship Between Patient Satisfaction After Cataract Surgery With Multifocal Intraocular Lens Implantation and Defocus Curves, Contrast Sensitivity and Photic Phenomena
Brief Title: Evaluating Patient Satisfaction After Cataract Surgery With Multifocal Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Clínica Rementería (Other)
Responsible Party: Sponsor
Other Study IDs: 18/552-E
Record Dates: First submitted 2018-12-23; First posted 2018-12-26 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Cataract
Keywords: Multifocal intraocular lens; Trifocal intraocular lens; Extended Depth of Focus Lens
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Cataract surgery — Evaluation of patient satisfaction after bilateral cataract surgery with multifocal intraocular lens implantation

SUMMARY:
Multifocal lens allow most patients to be spectacle-free after cataract surgery. Most studies published up-to-date have focused on visual acuity, but not on patient-reported outcomes. Since some patients with very good postoperative visual acuity report being very uncomfortable after surgery, the aim of this study is to evaluate if patient satisfaction is correlated with other outcomes, such as low-contrast visual acuity, contrast sensitivity, photic phenomena and ability to tolerate defocus. Patients who have undergone surgery with bilateral multifocal intraocular lens implantation will be carefully evaluated 3 months after surgery to try to determine the factors that correlate with patient reported outcomes as evaluated with the Catquest SF-9 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Previous bilateral cataract surgery
* Bilateral implantation of multifocal intraocular lens

Exclusion Criteria:

* Presence of ocular pathologies
* Intra- or postoperative complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone bilateral cataract surgery with bilateral implantation of a multifocal intraocular lens and who are willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | Three months after surgery
  Patient satisfaction with visual outcome three months after surgery as evaluated with the Catquest-9 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Inés Contreras, Principal Investigator — Clinina Rementería
Locations (1):
- Clínica Rementería, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rementeria-Capelo LA, Contreras I, Garcia-Perez JL, Carrillo V, Gros-Otero J, Ruiz-Alcocer J. Tolerance to Residual Refractive Errors After Trifocal and Trifocal Toric Intraocular Lens Implantation. Eye Contact Lens. 2021 Apr 1;47(4):213-218. doi: 10.1097/ICL.0000000000000726. PMID 33323876